CLINICAL TRIAL: NCT03595657
Title: A Single-Arm, Multicenter, Phase II Clinical Trial of CS1001 in Subjects With Relapsed or Refractory Extranodal Natural Killer/ T Cell Lymphoma(ENKTL)
Brief Title: A Study of CS1001 in Subjects With Relapsed or Refractory Extranodal Natural Killer/ T Cell Lymphoma(ENKTL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1001-201; CTR20180519 (Other: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Extranodal Natural Killer/T-Cell Lymphoma
Keywords: ENKTL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CS1001 (Experimental): Participants will receive CS1001 1200 mg by intravenous infusion every 3 weeks
  Interventions: Biological: CS1001

INTERVENTIONS:
Biological: CS1001 — monoclonal antibody

SUMMARY:
This is a multicenter, single-arm, phase II study to evaluate the efficacy and safety of CS1001 monotherapy for Relapsed or Refractory Extranodal Natural Killer/ T Cell Lymphoma (ENKTL)

DETAILED DESCRIPTION:
Eligible subjects with rr-NKTL after prior asparaginase-based chemotherapy or chemo radiotherapy are planned to receive CS1001 1200 mg intravenous infusion every three weeks until progression of disease, intolerable toxicity, consent withdrawn, death. The primary endpoint of this trial is objective response rate (ORR), as assessed by independent radiological review committee (IRRC) based on Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a histologically confirmed NKTL at study site.
2. Subject must have relapsed or refractory NKTL after prior asparaginase-based chemotherapy or chemo radiotherapy.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
4. Subject must have at least one evaluable or measurable lesion per Lugano 2014 classification.
5. Subject must have adequate organ function and bone marrow function without severe hematopoietic disorder, or heart, lung, liver or kidney dysfunction or immune deficiency.
6. Subject must provide stained tumor tissue sections and corresponding pathological report or unstained tumor tissue sections (or tissue block) for central pathology review.
7. Subject with prior anti-cancer treatment can only be enrolled when the toxicity of prior anti-cancer treatment has recovered to baseline or ≤ Grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

Exclusion Criteria:

1. Invasive natural killer leukemia.
2. Concomitant with hemophagocytic syndrome.
3. Primary site in central nervous system (CNS) or CNS involvement.
4. Subjects currently participating in other clinical studies or use of any investigational drug within 4 weeks prior to the first dose of CS1001.
5. Subjects who received systemic corticosteroid or any other immunosuppressive therapy within 14 days prior to the first dose of CS1001.
6. Subjects who had prior chemotherapy, immune therapy, biological therapy as systemic treatment for cancer, within 28 days prior to the first dose of CS1001.
7. Receipt of traditional medicinal herbal preparations with anti-tumor indications with 7 days prior to the first dose of CS1001.
8. Known history of human immunodeficiency virus (HIV) infection and/or acquired immune deficiency syndrome.
9. Subjects with active hepatitis B or C infection.
10. Subjects with active tuberculosis infection.
11. Subjects who received prior therapy with anti-PD-1, anti-PD-L1 or anti-CTLA-4 monoclonal antibody.
12. Female subjects who are pregnant or breast-feeding.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Peking University Third Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen University Cancer Prevention Center, Guangzhou
  - Guizhou Cancer Hospital, Guiyang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Cancer Hospital, Hefei
  - Cancer Hospital Affiliated to Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - Cancer Center of Union Hospital, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou

REFERENCES:
- [Derived] Huang H, Tao R, Hao S, Yang Y, Cen H, Zhou H, Guo Y, Zou L, Cao J, Huang Y, Jin J, Zhang L, Yang H, Xing X, Zhang H, Liu Y, Ding K, Qi Q, Zhu X, Zhu D, Wang S, Fang T, Dai H, Shi Q, Yang J. Sugemalimab Monotherapy for Patients With Relapsed or Refractory Extranodal Natural Killer/T-Cell Lymphoma (GEMSTONE-201): Results From a Single-Arm, Multicenter, Phase II Study. J Clin Oncol. 2023 Jun 1;41(16):3032-3041. doi: 10.1200/JCO.22.02367. Epub 2023 Mar 30. PMID 36996373

RESULTS

PARTICIPANT FLOW:
Groups:
- R/R ENKTL: Participants received sugemalimab (CS1001) 1200 mg intravenously every 3 weeks (Q3W)
Period: Overall Study
Arm/Group | R/R ENKTL
Started | 80
Completed | 13
Not Completed | 67
Not completed — Adverse Event | 14
Not completed — Death | 1
Not completed — Lack of Efficacy | 40
Not completed — Withdrawal by Subject | 10
Not completed — Dosing delayed over 9 weeks | 1
Not completed — Achieved CR and completed 2 years of treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 80
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 80
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — 0-Fully active, able to carry on all pre-disease performance without restriction. 1-Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. 2-Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. 3-Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. 4-Completely disabled; cannot carry on any selfcare; totally confined to bed or chair. 5-Dead
  Participants
    0 | 21
    1 | 59
Stage of Extranodal Natural Killer/ T-cell Lymphoma at screening [Count of Participants; unit: Participants] — Based on Ann Arbor classification: Stage I - Involvement: 1 node or a group of adjacent nodes. Extranodal Status: Single extranodal lesion without nodal involvement. Stage II - Involvement: 2 or more nodal groups on the same side of the diaphragm. Extranodal Status: Stage I/II by nodal extent with limited contiguous extranodal involvement. Stage III - Involvement: Nodes on both sides of the diaphragm; nodes above the diaphragm with spleen involvement. Extranodal Status: N/A. Stage IV - Involvement: Additional noncontiguous extralymphatic involvement. Extranodal Status: N/A.
  Participants
    Stage I | 9
    Stage II | 17
    Stage IV | 54
Epstein-Barr Virus (EBV) DNA at Screening [Count of Participants; unit: Participants]
  Positive | 44
  Negative | 36
Baseline Bone Marrow Assessment Result [Count of Participants; unit: Participants] — Assessments were performed at baseline to determine whether a patient had bone marrow involvement by the disease. "Positive" indicates the presence of involvement; "negative" indicates absence of involvement; "missing" indicates results not applicable.
  Participants
    Positive | 5
    Negative | 73
    Missing | 2
Central Pathology Confirmed ENKTL [Count of Participants; unit: Participants]
  Yes | 79
  No | 1
Patient Status [Count of Participants; unit: Participants] — Participants in this study must have relapsed or refractory ENKTL failing asparaginase-based chemotherapy or chemoradiotherapy. "Relapse" indicates disease progression after response to the last treatment; "refractory" indicates no response to the last treatment.
  Participants
    Relapsed | 43
    Refractory | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assessed by IRRC
Description: ORR assessed by the independent radiological review committee (IRRC) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: Two patients were excluded from analysis: one patient was not confirmed as ENKTL by central pathology, and the other patient was identified as having no measurable or evaluable disease at baseline by IRRC.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 78
percentage of Participants | 46.2 [34.8 to 57.8]

2. Secondary Outcome: Objective Response Rate (ORR) Assessed by Investigators
Description: ORR assessed by investigators according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: One patient was excluded from the efficacy analysis set because the patient was not confirmed as ENKTL by central pathology.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
Percentage of participants | 45.6 [34.3 to 57.2]

3. Secondary Outcome: Complete Response Rate (CRR) by Investigators
Description: CRR assessed by investigators according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
Percentage of participants | 30.4 [20.5 to 41.8]

4. Secondary Outcome: Complete Response Rate (CRR) Assessed by IRRC
Description: CRR assessed by the independent radiological review committee (IRRC) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 78
Percentage of participants | 37.2 [26.5 to 48.9]

5. Secondary Outcome: Partial Response Rate (PRR) Assessed by Investigators
Description: PRR assessed by the investigators according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
Percentage of participants | 15.2 [8.1 to 25.0]

6. Secondary Outcome: Partial Response Rate (PRR) Assessed by IRRC
Description: PRR assessed by the independent radiological review committee (IRRC) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 78
Percentage of participants | 9.0 [3.7 to 17.6]

7. Secondary Outcome: Duration of Response (DoR) Assessed by Investigators
Description: DoR assessed by the investigators according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
months | 39.9 [14.8 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

8. Secondary Outcome: Duration of Response (DoR) Assessed by IRRC
Description: DoR assessed by the independent radiological review committee (IRRC) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 78
months | 35.2 [25.3 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

9. Secondary Outcome: Time to Response (TTR) Assessed by Investigators
Description: TTR assessed by the investigators according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
months | 2.8 [1.4 to 8.0]

10. Secondary Outcome: Time to Response (TTR) Assessed by IRRC
Description: TTR assessed by the independent radiological review committee (IRRC) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: From enrollment to end of follow-up, a median of 29 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 78
months | 2.8 [1.4 to 11.1]

11. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: From enrollment to end of follow-up, a median of 29 months
Measure: Count of Participants; unit: Participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 80
Participants
  Treatment-Emergent Adverse Event (TEAE) | 77
  Treatment-Related Adverse Event (TRAE) | 63
  Serious Adverse Event (SAE) | 22
  Related SAE | 8
  ≥G3 TEAE | 37
  ≥G3 TRAE | 15
  Infusion-related Reaction | 4
  TEAE of special interest | 24
  TEAE of special interest grade 3-5 | 2
  TEAE Leading to Death | 5
  TEAE Leading to Drug Permanently Discontinued | 14
  TEAE Leading to Infusion Interruption | 4
  TEAE Leading to Treatment Cycle Delay | 22

12. Other Pre Specified Outcome: 6-months Progression-free Survival (PFS) Rate Assessed by Investigators
Description: 6-months PFS rate assessed by the investigators according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
Percentage of participants | 39.1 [28.1 to 49.9]

13. Other Pre Specified Outcome: 6-months PFS Rate Assessed by IRRC
Description: 6-months PFS rate assessed by the independent radiological review committee (IRRC) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 78
percentage of participants | 49.7 [38.0 to 60.3]

14. Other Pre Specified Outcome: 6-month Overall Survival (OS) Rate
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R/R ENKTL
Number analyzed (Participants) | 79
Percentage of participants | 79.2 [68.3 to 86.7]

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, a median of 29 months
Arm/Group | R/R ENKTL
All-Cause Mortality (participants affected / at risk) | 37/80
Serious Adverse Events (participants affected / at risk) | 22/80
Other Adverse Events (participants affected / at risk) | 76/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R/R ENKTL (N=80)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Deafness bilateral (Ear and labyrinth disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Pyrexia (General disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2
Fungaemia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Septic shock (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Ear injury (Injury, poisoning and procedural complications) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R/R ENKTL (N=80)
Anaemia (Blood and lymphatic system disorders) | 14
Hyperthyroidism (Endocrine disorders) | 5
Hypothyroidism (Endocrine disorders) | 18
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 25
COVID-19 (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 21
Blood bilirubin increased (Investigations) | 6
Blood creatinine increased (Investigations) | 4
Blood thyroid stimulating hormone decreased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 10
Haemoglobin decreased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 13
Neutrophil count decreased (Investigations) | 21
Platelet count decreased (Investigations) | 11
Protein urine present (Investigations) | 8
Thyroxine free decreased (Investigations) | 6
Urinary occult blood positive (Investigations) | 6
Urobilinogen urine increased (Investigations) | 4
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 25
White blood cells urine positive (Investigations) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypochloraemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Hypoaesthesia (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the sponsor has not published trial results within 18 months since trial completion, the PI is allowed to publish data collected at the corresponding site. The PI should provide draft publication to the sponsor to review prior to distribution to any external parties; the sponsor should provide review comments to the PI within 60 calendar days since receipt of draft publication; the sponsor also has rights to postpone publication for up to 6 months based on reasonable grounds.

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03595657/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT03595657/SAP_001.pdf